CLINICAL TRIAL: NCT06489808
Title: An Open-label, Multicenter, Multi-cohort Clinical Study of Linperlisib Combined With Standard Immunochemotherapy in the Treatment of Relapsed/Refractory Large B-Cell Lymphoma Failing to First-line Therapy
Brief Title: Linperlisib Combined With Immunochemotherapy in Relapsed/Refractory LBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024030
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: Relapsed/Refractory Large B-Cell Lymphoma
Keywords: Linperlisib; Immunochemotherapy
MeSH Terms: conditions — Recurrence | interventions — Rituximab; Gemcitabine; Oxaliplatin; Ifosfamide; Carboplatin; Etoposide; Dexamethasone; Cisplatin; Cytarabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 transplant-ineligible patients: Linperlisib combined with R-Gemox regimen (Experimental): Cohort 1 consisted of transplant-ineligible patients who received Linperlisib in combination with R-Gemox. The treatment regimen was as follows: Linperlisib (RP2D dosage) on Days 1-14, rituximab 375 mg/m² on Day 0, gemcitabine 1000 mg/m² on Day 1, and oxaliplatin 130 mg/m² on Day 1, every 21 days for 6 cycles.
  Interventions: Drug: Linperlisib; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin
- Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens (Experimental): Cohort 2 consisted of patients scheduled for transplantation who received 3 cycles of Linperlisib (RP2D, D1-14) combined with R-ICE/DHAP/GVM regimen (R-ICE regimen: rituximab, ifosfamide, carboplatin, etoposide; R-DHAP regimen: rituximab, cytarabine, dexamethasone, cisplatin; R-GVM regimen: rituximab, gemcitabine, vinorelbine, mitoxantrone liposome), followed by autologous hematopoietic stem cell transplantation in responding patients.
  Interventions: Drug: Linperlisib; Drug: Rituximab; Drug: Gemcitabine; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Dexamethasone; Drug: Cisplatin; Drug: Ara-C; Drug: Vinorelbine; Drug: Mitoxantrone hydrochloride liposome

INTERVENTIONS:
Drug: Linperlisib — Linperlisib RP2D D1-14
Drug: Rituximab — rituximab 375 mg/m2 D0
Drug: Gemcitabine — gemcitabine per regimen dosage
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 D1
  Arms: Cohort 1 transplant-ineligible patients: Linperlisib combined with R-Gemox regimen
Drug: Ifosfamide — Ifosfamide 5g/m2 D2
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Carboplatin — Carboplatin AUC=5mg/mL · min (maximum absolute dose/cycle = 800 mg)
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Etoposide — Etoposide 100mg/m2 D1-3
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Dexamethasone — Dexamethasone 40mg D1-4
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Cisplatin — Cisplatin 100mg/m2 D1, continuous intravenous infusion
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Ara-C — Ara-C 2g/m2 q12h D2
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Vinorelbine — Vinorelbine 20mg/m2 D1
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens
Drug: Mitoxantrone hydrochloride liposome — Mitoxantrone hydrochloride liposome 18mg/m2 D1
  Arms: Cohort 2 patients scheduled for transplantation:Linperlisib combined with R-ICE/DHAP/GVM regimens

SUMMARY:
To evaluate the efficacy and safety of Linperlisib combined with standard immunochemotherapy in patients with R/R LBCL.

DETAILED DESCRIPTION:
This is a phase 2, open-label, multicenter, multi-cohort study evaluating the efficacy and safety of Linperlisib combined with standard immunochemotherapy in the treatment of relapsed/refractory LBCL after first-line treatment. This study is divided into a safety run-in phase and a dose expansion phase.The primary objective of the safety run-in phase was to determine the recommended dose for the dose expansion phase based on dose-limiting toxicities (DLTs).

The dose expansion phase consisted of Cohort 1 and Cohort 2.Cohort 1 was transplant-ineligible patients who received Linperlisib in combination with R-Gemox at RP2D for 6 cycles.Cohort 2 consisted of patients scheduled for transplantation who received 3 cycles of Linperlisib combined with R-ICE/DHAP/GVM regimen, followed by autologous hematopoietic stem cell transplantation in responding patients

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed large B-cell lymphoma (LBCL), including diffuse large B-cell lymphoma unspecified (DLBCL, NOS), follicular lymphoma grade 3B (FL, 3B), high-grade B-cell lymphoma unspecified (HGBCL, NOS), DLBCL/HGBCL with MYC and BCL2 rearrangements, FL transformed DLBCL without a previous history of indolent lymphoma.
2. Relapsed or refractory after first-line immunochemotherapy (which must include CD20 monoclonal antibody and anthracycline) 1)Refractory is defined as failure to achieve a complete response to first-line therapy (excluding patients who are intolerant to first-line therapy), including progressive disease (PD) as the best response to first-line therapy; stable disease (SD) as the best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R-CHOP); partial response (PR) as the best response after at least 6 cycles of first-line therapy with biopsy-confirmed residual disease or disease progression within 12 months of initiating first-line therapy; complete response to first-line therapy followed by progression within 12 months after the end of therapy. 2)Relapse was defined as a complete response to first-line therapy followed by progression confirmed more than 12 months after the end of therapy.
3. Subjects must have at least 1 measurable lesion/evaluable lesion that meets the 2014 version of the Lugano Lymphoma Evaluation Criteria.
4. Subjects has no known or suspected central nervous system involvement by lymphoma.
5. Previous treatment with any antineoplastic therapy (including radiation therapy, chemotherapy, hormonal therapy, surgery, or molecular targeted therapy) for which participation in this trial must have exceeded 2 weeks or 5 drug half-lives, whichever is shorter.
6. Age ≥ 18 years.
7. ECOG score 0-2.
8. Expected survival ≥ 3 months.
9. Women of Childbearing Potential subjects must have a negative serum/urine pregnancy test within 7 days prior to the first dose; female subjects of childbearing potential and male subjects with partners of childbearing potential, as well as their partners, should agree to use effective contraception from signing the ICF until 6 months after the last dose of study drug.
10. Able to comply with the trial protocol as judged by the investigator.
11. Each subject (or legally acceptable representative) voluntarily joined the study and signed an informed consent form.

    -

Exclusion Criteria:

1. Other malignancies within the last 5 years, except radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the breast, and carcinoma in situ of the cervix.
2. Previous autologous or allogeneic hematopoietic stem cell transplantation.
3. History of Richter transformation.
4. Received > 1 line of systemic antineoplastic therapy.
5. Prior treatment with PI3K inhibitors.
6. Known hypersensitivity to trial products.
7. Active viral, bacterial, or fungal infection requiring treatment (eg, pneumonia, etc.).
8. Requiring prolonged systemic hormones (at doses equivalent to > 10 mg prednisone/day) or any other form of immunosuppressive therapy. Subjects taking inhaled or topical corticosteroids may be enrolled.
9. Concomitant diseases and medical history:

   1. Multiple factors affecting oral medication (e.g. inability to swallow, chronic diarrhea, ileus, etc.).
   2. Patients with a history of psychotropic substance abuse who cannot quit or have mental disorders.
   3. Subjects with any severe and/or uncontrolled disease including:

      1)Unsatisfactory blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg). 2)Patients with ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 450 ms (male), QTc ≥ 470 ms (female)) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification). 3)Active interstitial pneumonia or other chronic lung disease resulting in severely impaired lung function defined as FEV1 and DLCOc < 60% of predicted normal; history of interstitial pneumonia due to COVID-19. 4)Abnormal liver: I.Decompensated cirrhosis (Child-Pugh class B or C). II.Known history of clinically significant liver disease. 5)Renal failure requiring hemodialysis or peritoneal dialysis. 6)Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage. 7)Urine routine showed urine protein ≥ + +, and confirmed 24-hour urine protein quantification > 1.0 g.
   4. Patients with active or history of autoimmune diseases that may relapse (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or patients at high risk. Patients with autoimmune hypothyroidism requiring only hormone replacement therapy may be considered for enrollment if the disease is stable as assessed by the investigator.
10. Known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome.
11. Positive pregnancy test at baseline in female patients who are pregnant, lactating, or of childbearing potential.
12. Concurrent medical conditions that, in the investigator 's judgment, would seriously compromise the patient' s safety or the patient 's completion of the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities | Safety Run-in Period, up to the end of cycle 1 (each cycle is 21 days)
  Dose-Limiting Toxicities per study protocol defination
ORR | up to 2 years
  Response is assessed according to the Lugano criteria

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 2 years
  The adverse events were evaluated by NCI-CTCAE 5.0 standard Hematologic and non-hematologic toxicity
Complete Response Rate (CRR) | up to 2 years
  Response is assessed according to the Lugano criteria
Duration of Response (DOR) | up to 2 years
  From the date of achieving complete or partial response until disease progression, death or last follow-up
Duration of Complete Response (DOCR) | up to 2 years
  From the date of achieving complete response until disease progression, death or last follow-up
Progression-free Survival (PFS) | up to 2 years
  From the date of the first dose of therapy is given until disease progression, death or last follow-up
Overall Survival (OS) | up to 2 years
  From the date of the first dose of therapy is given until death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, CAMS & PUMC
Locations (1):
- Institute of Hematology & Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No